CLINICAL TRIAL: NCT04047290
Title: A Phase 1a/1b, Multicenter, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK112 in Subjects With Advanced Solid Tumors
Brief Title: A Study of AK112, a PD-1/VEGF Bispecific Antibody, for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK112-101
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Neoplasms Malignant
Keywords: anti-PD-1/VEGF bispecific antibody; immunotherapy; immuno-oncology; advanced solid tumors; bispecific; PD-1/VEGF
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Initially, a single-subject cohort will be enrolled at the protocol starting dose of AK112 every 2 weeks (Q2W). Dose escalation will proceed to the next main dose level according to the 3+3+3 dose-escalation procedure until the MTD is reached. Dose expansion phase of the study will be initiated at the Sponsor's discretion at the dose level and treatment schedule which was established as the recommended Phase 2 dose (RP2D) in the dose-escalation phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AK112 (Experimental): AK112 IV every 2 weeks (q2w) or every 3 weeks (q3w)
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — AK112 is a PD1/VEGF bispecific antibody.

SUMMARY:
This study is to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of AK112, a PD-1/VEGF bispecific antibody, as a single agent in adult subjects with advanced solid tumor malignancies. The study consists of a dose escalation phase (Phase 1a) to determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for AK112 as a single agent, and a dose expansion phase (Phase 1b) in subjects with specific tumor types which will characterize treatment of AK112 as a single agent at the MTD or RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent and any locally required authorization obtained from the subject/legal representative.
* In dose-escalation cohorts (Phase 1a), histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject refuses standard therapy.
* In the dose-expansion cohorts (Phase 1b), histologically or cytologically confirmed selected advanced solid tumors.
* Subject must have at least one measurable lesion according to RECIST Version1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
* Available archived tumor tissue sample to allow for correlative biomarker studies. If unavailable or unsuitable, the subject must consent and undergo fresh tumor biopsy.
* Adequate organ function.
* Subjects with central nervous system (CNS) metastases must have been treated, be asymptomatic.
* Females of childbearing potential and non-sterilized males who are sexually active must use an effective method of contraception from screening until 120 days after final dose of investigational product or women of non child bearing potential.
* Life expectancy ≥12 weeks.

Exclusion Criteria:

* History of severe hypersensitivity reactions to other mAbs.
* Prior malignancy active within the previous 3 years except for the tumor for which a subject is enrolled in the study, and locally curable cancers that have been apparently cured, (e.g. basal cell skin cancer, or carcinoma in situ of the cervix or breast).
* For subjects enrolled in the dose escalation phase, having received prior anti-PD-1, anti-PD-L1, anti-CTLA-4 or any other immunotherapy or immune-oncology (IO) agent within 28 days of commencing treatment with AK112 or experienced a toxicity that led to permanent discontinuation of prior immunotherapy. All AEs while receiving prior immunotherapy have not completely resolved or resolved to Grade 1 prior to screening, required the use of additional immunosuppression other than corticosteroids
* Receiving any immunotherapy, conventional or investigational systemic anticancer therapy within 4 weeks prior to the first dose
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment (hormones use for non-cancer related conditions is acceptable).
* Subjects with clinically significant cardiovascular disease
* Subjects with a condition requiring systemic treatment with either corticosteroid (> 10 mg daily ) or other immunosuppressive medications within 2 weeks of study drug administration.
* Current or recent use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
* Current unstable of full-dose oral or parenteral anticoagulants or thrombolytic agents for > 2 weeks prior to the first dose of AK112
* Active or prior documented autoimmune disease within the past 2 years or conditions not expected to recur in the absence of an external trigger)
* Active or prior documented inflammatory bowel disease
* History of primary immunodeficiency.
* History of organ transplant.
* Known allergy or reaction to any component of the AK112 formulation.
* History of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1
* Major surgical procedure within 30 days prior to the first dose of AK112 or still recovering from prior surgery.
* Known history of HIV.
* Known active hepatitis B or C infections. Note: Subjects with HCC and positive HBsAg result are eligible if the subjects were treated with antiviral therapy and HBV viral load less than 500 IU/mL prior to first dose of AK112.
* An active infection requiring systemic therapy
* Received live attenuated vaccination within 30 days prior to the first dose of AK112.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of participants with adverse events (AEs) | From time ICF is signed until 90 days after last dose of AK112
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with DLTs | During the first four weeks of treatment with AK112
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle (4 weeks) of treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD at 16 and 24 weeks respectively) based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK112 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with AK112 until death due to any cause.
Area under the curve (AUC) of AK112 for assessment of pharmacokinetics | From first dose of AK112 through 90 days after last dose of AK112
  The endpoints for assessment of PK of AK112 include serum concentrations of AK112 at different timepoints after AK112 administration.
Maximum observed concentration (Cmax) and Minimum observed concentration (Cmin) of AK112 | From first dose of AK112 through 90 days after last dose of AK112
  The endpoints for assessment of PK of AK112 include serum concentrations of AK112 at different timepoints after AK112 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK112 through 90 days after last dose of AK112
  The immunogenicity of AK112 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Border Medical Oncology, Albury, New South Wales
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - ICON Cancer Foundation, South Brisbane, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frentzas S, Austria Mislang AR, Lemech C, Nagrial A, Underhill C, Wang W, Wang ZM, Li B, Xia Y, Coward JIG. Phase 1a dose escalation study of ivonescimab (AK112/SMT112), an anti-PD-1/VEGF-A bispecific antibody, in patients with advanced solid tumors. J Immunother Cancer. 2024 Apr 19;12(4):e008037. doi: 10.1136/jitc-2023-008037. PMID 38642937
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38642937/